CLINICAL TRIAL: NCT05439642
Title: Validation and Reliability of the Canadian Haemophilia Outcomes-Kids' Life Assessment Tool (CHO-KLAT) in Turkish
Brief Title: Validation and Reliability of the CHO-KLAT in Turkish
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuzuncu Yil University (Other)
Collaborators: Hasan Kalyoncu University (Other); University of Gaziantep (Other); Acıbadem Adana Hospital (Other)
Responsible Party: Principal Investigator, Ayse Merve TAT, Assistant Professor, Yuzuncu Yil University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: YuzuncuYıl2022/1
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Hemophilia; Health Related Quality of life
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Intervention Model Description: Validation and reliability study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemophilia (Other): Evaluation of quality of life of children with hemophilia in Turkey
  Interventions: Other: Evaluation of health related quality of life

INTERVENTIONS:
Other: Evaluation of health related quality of life — Evaluation of health related quality of life of boys with hemophilia with the Canadian Haemophilia Outcomes-Kids' Life Assessment Tool and the Pediatric Inventory of Quality of Life

SUMMARY:
The aim of this study is to investigate the Turkish validity and reliability of the Canadian Haemophilia Outcomes-Kids' Life Assessment Tool version2.0. Patients aged 4-18 years with hemophilia a or b will be included in the study. The study was planned as a multicenter and it is aimed to reach 100 patients. The process included four steps: a linguistic adaptation, cognitive debriefing interviews with children and their parents, a validity assessment with the Pediatric Quality of Life Inventory (PedsQL) as a comparator, and a test retest reliability assessment.

DETAILED DESCRIPTION:
Health-related quality of life assessment is considered an important outcome in the evaluation of children with hemophilia. The Canadian Haemophilia Outcomes-Kids' Life Assessment Tool version2.0 is a disease-specific health-related quality of life measurement tool for 4 to 18-year-old boys with haemophilia. The aim of this study is to ensure the use of CHO-KLAT in clinical studies in Turkey.

Methods: Patients aged 4-18 years with hemophilia a or b will be included in the study.The study will be carried out in Van, Gaziantep and Adana provinces in Turkey and and it is aimed to reach 100 patients with hemophilia. The process included four steps: a linguistic adaptation, cognitive debriefing interviews with children and their parents, a validity assessment with the Pediatric Quality of Life Inventory (PedsQL) as a comparator, and a test retest reliability assessment.

ELIGIBILITY:
Inclusion Criteria:

* have Hemophilia A or B

Exclusion Criteria:

* Did not have significant cognitive impairment

Ages: 4 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
HRQoL questionnaire | 1-2 week
  Health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Merve Tat, Asst.Prof, Study Director — Van Yuzuncu Yıl University Faculty of Health Sciences; Tugba Badat Gonen, PhD, Principal Investigator — Hasan Kalyoncu University Faculty Of Health Sciences; Ahmet Fayik Oner, Prof MD, Study Chair — Van Yuzuncu Yıl University Faculty of Medicine
Locations (4):
- Turkey (Türkiye) (4):
  - Adana Acibadem Hospital, Adana
  - Gaziantep University, Gaziantep
  - Hasan Kalyoncu University, Gaziantep
  - Van Yuzuncu Yıl University, Van